CLINICAL TRIAL: NCT06323512
Title: Pulmonary Artery Denervation for Treatment of Patients With Heart Failure Without Pulmonary Hypertension: a Safety and Proof-of-principle Cohort Study
Brief Title: Pulmonary Arteyr Denervation for HF Without PH
Status: Completed | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shaoliang Chen, MD, Professor, Nanjing First Hospital, Nanjing Medical University
Other Study IDs: Nanjing
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Pulmonary artery denervation (PADN) — Combining invasive angiography with pulmonary artery CTA is frequently employed to determine the final size of the PADN catheter, aiming for an expected ratio of distal ring/vessel diameter between 1.1 and 1.2. The PADN system comprises a radiofrequency generator, connecting tubing and control handle, and the PADN catheter. The main interface of the radiofrequency generator offers multiple language options and displays parameters such as temperature, impedance, energy, and ablation time. The generator features three control modes: temperature control, power control, and a combination of both.

SUMMARY:
Prolonged pulmonary venous congestion culminates in pulmonary hypertension, defined as a mean pulmonary arterial pressure > 20 mmHg and pulmonary artery wedge pressure >15 mmHg at rest, as determined by right heart catheterization. Pulmonary hypertension secondary to heart failure (PH-HF) is further stratified into isolated post-capillary pulmonary hypertension (Ipc-PH, pulmonary vascular resistance (PVR) is ≤2 Woods Unit) and combined pre- and post-capillary pulmonary hypertension (Cpc-PH, PVR > 2 Woods Unit), the later reflecting additional pulmonary vascular constriction or remodeling in addition to passive PH. While medications tailored for World Health Organization defined Group I pulmonary arterial hypertension are not endorsed for PH-HF according to current guidelines, the coexistence of pulmonary hypertension exacerbates the severity of heart failure. Given the presence of pulmonary arterial vasoconstrictor and heightened sympathetic nervous activity in patients with heart failure, the PADN-5 study has demonstrated the safety and efficacy of pulmonary artery denervation (PADN) for patients with CpcPH, characterized by the improvements in left ventricular ejection fraction, cardiac output, clinical outcome, and reductions in left atrial pressure, pulmonary arterial pressure, and PVR. Our objective is to assess the feasibility, safety, and efficacy of PADN for patients with heart failure independent of left ventricular ejection fraction (HFrEF or HFpEF) without pulmonary hypertension (N=30, 15 with HFrEF and another 15 with HFpEF).

DETAILED DESCRIPTION:
We conducted a safety and proof-of-principle cohort study at a single centre in China. Eligible patients, aged 18 years or greater, had a documented history of chronic (≥6 months) ischaemic or non-ischaemic cardiomyopathy. They also met the American College of Cardiology/American Heart Association (ACC/AHA) stage C heart failure criteria, with New York Heart Association (NYHA) class III or ambulatory class IV symptoms. Additionally, participants were required to have been receiving guideline-directed medical therapy for at least three months, as tolerated per ACC/AHA guidelines.

Further inclusion criteria encompassed a pulmonary artery wedge pressure exceeding 15 mm Hg, a mean pulmonary arterial pressure less than or equal to 20 mm Hg, and pulmonary vascular resistance (PVR) less than or equal to 2 Woods Unit. Patients were ineligible if they lacked patent femoral venous or inferior vena cava/right jugular vein access, or exhibited a plasma N-terminal prohormone B-type natriuretic peptide (NT-proBNP) level below 300 pg/ml, had experienced a stroke or thromboembolic event within the preceding 12 months, had patent foramen ovale or atrial septal defect, or presented with severe (grade 4) mitral regurgitation. Patients with coagulation disorders or contraindications for oral anticoagulation, as well as those harboring pulmonary artery, right atrial, or right ventricular thrombus, were also excluded.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or greater, had a documented history of chronic (≥6 months) ischaemic or non-ischaemic cardiomyopathy; ACC/AHA stage C heart failure criteria, NYHA class III or ambulatory class IV symptoms; on GDMT for heart failure at least three months; PAWP exceeding 15 mm Hg, mean PAP less than or equal to 20 mm Hg, and PVR less than or equal to 2 Woods Unit

Exclusion Criteria:

Patients lacked patent femoral venous or inferior vena cava/right jugular vein access; had experienced a stroke or thromboembolic event within the preceding 12 months, had patent foramen ovale or atrial septal defect, or presented with severe (grade 4) mitral regurgitation; had coagulation disorders or contraindications for oral anticoagulation; had harboring pulmonary artery, right atrial or right ventricular thrombus; had undergone pacemaker implantation within 1 month.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Left ventricular dp/dt (maximal and minimal) | before and immediately after PADN procedures
Left ventricular end-systolic pressure (maximal and minimal) | Before and immediately after PADN procedures

SECONDARY OUTCOMES:
Pulmonary arterial wedge pressure | Before, after-PADN and at 3 months
  PAWP
Tricuspid annuls peak systolic excursion | Before, after-PADN and at 3 months
  TAPSE
NT-proBNP | Before, after-PADN and at 3 months
  N-terminal-pro brain natriuretic peptide

CONTACTS AND LOCATIONS:
Overall Officials: Hongjuan C Peng, MBBS, Study Director — Nanjing First Hospital, Nanjing Medical University, China
Locations (1):
- Nanjing First Hospital, Nanjing, Please Select, China

IPD SHARING:
Plan to Share IPD: Undecided